CLINICAL TRIAL: NCT05836194
Title: Comparison of Ultra-Widefield Scanning Laser Ophthalmoscopy and Two-Field Fundus Photography for Evaluating Diabetic Retinopathy
Brief Title: Evaluation of Diabetic Retinopathy Using Ultra-Widefield Fundus Images Compared With Two-Field Fundus Images
Status: Completed | Type: Observational
Sponsor: Ningbo Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DRUWFVSFP20230501
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Retinal Diseases; Diabetic Retinopathy; Diabetes Complications; Diabetes Mellitus; Screening
Keywords: Diabetic Retinopathy; Ultra wide-field imaging; Fundus Photography; Screening
MeSH Terms: conditions — Retinal Diseases; Diabetic Retinopathy; Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the accuracy of evaluating diabetic retinopathy using ultra-widefield fundus images versus two-field fundus images. The hypothesis is that screening and grading diabetic retinopathy based on ultra-widefield fundus images may yield higher accuracy compared to the use of two-field fundus images.

DETAILED DESCRIPTION:
As of 2030,9.7% (108.4 million) people in the China population have diabetes, and the total costs of diabetes in adults would reach $460.4 billion. Diabetic retinopathy (DR) and diabetic macular oedema (DME) are the principal causes of adult vision loss. Nevertheless,DR has few visual symptoms until DME occurs or the lessions located in the peripheral retina.Thus,it is crucial to early diagnosis and treatment of DR patients,which will prevent vision loss and reduce the societal buren of diabetes.

The Early Treatment Diabetic Retinopathy Study (ETDRS) standard 7-field 30° color fundus photography is a time-consuming examination requiring pharmacological pupil dilation,experienced photographers and image montage.To simplify the operation process and improve patient compliance,2-field 45° retinal photographs (1 macular-centered field and 1 disc-centerde field) was proposed in the EURODIAB IDDM complications study and widely used in DR screening.Two-field 45° retinal photographs has been proven beneficial in reducing blindness resulting from DR,while may be neglected DR pathology in the peripheral retina.With the development of imaging technology, nonmydriatic ultra-widefield scanning laser opthoalmascopy (optomap) can obtain high-resolution,widefield images (180-200°) of the retina in only 0.25s. Optomap had good agreement with 7-field ETDRS in determining DR and DME severity and may be profitable in DR evaluation in research and clinical settings,espesially in predominantly peripheral lession(PPL).

Patients with DM, with or without known DR, will be imaged using the optomap and 2-field 45° retinal photographs imaging device both for diagnosis and screening purposes at Ningbo Eye Hospital. Internal validation and continuous quality control will routinely be conducted. According to the International Clinical Diabetic Retinopathy Disease Severity Scale, the data for the ungradable image rate, distribution of DR severity levels, and PPL will be evaluated and compared. Statistics analysis will explore the agreement of DR severity levels between optomap images and 2-field photographs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of diabetes mellitus.

Exclusion Criteria:

1. Diseases involving the posterior pole other than DR, such as age-related macular degeneration，retinal vein occlusion.
2. History of panretinal laser photocoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18 and older) with diabetes presenting at the outpatient clinic of the Department of Ophthalmology, Ningbo Eye Hospital, practice for examination of diabetic retinopathy.
Sampling Method: Non-Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The International Clinical Diabetic Retinopathy Disease Severity Scale within the 2-fields fundus photography and Ultra-Wide field scanning laser ophthalmoscopy (Optomap) imaging and statistical comparison | 60 days
  To compare nonmydriatic 2-fields fundus photographs with nonmydriatic ultra-wide field images for determining diabetic retinopathy(DR) severity. DR severity level agreement will be cross-tabulated, and Kappa value will be calculated.

SECONDARY OUTCOMES:
Number of Ungradable Images within the 2-field fundus photography and Optomap imaging | 7 day
  The proportion and reasons of ungradable images will be documented.
Number of predominantly peripheral lession(PPL) with Optomap imaging | 7 day
  The proportion of PPL images will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotian Liu, MD, Study Director — Ningbo Eye Hospital
Locations (1):
- Ningbo Eye Hospital, Ningbo, Zhejiang, China